CLINICAL TRIAL: NCT06360432
Title: Effects of the EatWelLog App on Enhancing Daily Diet Management for Community-dwelling Older Adults With Sarcopenic Obesity: A Pilot Randomized Controlled Trial
Brief Title: Effects of the EatWelLog App on Diet Management for Older Adults With Sarcopenic Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240214001
Record Dates: First submitted 2024-03-20; First posted 2024-04-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic Obesity; m-health; dietary intervention; exercise; behaviour change
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A two-arm, assessor-blinded, parallel design pilot randomized control trial (RCT) consisting of a M-health and a control group will be adopted to evaluate the effectiveness of the EatWellLog App in improving older adults' sarcopenic obesity (SO) status and other SO-related parameters by enhancing the self-management abilities and longer-term adherence to daily diet management among participants in the M-health group using the App, compared to the control group.
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is blinded to the group allocations will assess the participants' outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-health group (Experimental): Participants in the M-health will receive an 8-week program consisting of personalized dietary modification program and group-based exercise training. Additionally, the m-health group will be instructed to use the EatWellLog app for daily diet self-management.
  Interventions: Behavioral: Dietary modification program; Behavioral: Exercise training; Behavioral: The EatWellLog App
- Control group (Sham Comparator): Participants in the Control group will receive an identical, 8-week program consisting of personalized dietary modification program and group-based exercise training without using the EatWellLog App.
  Interventions: Behavioral: Dietary modification program; Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Dietary modification program — Participants will receive an 8-week program consisting of personalized dietary modification program. The dietary modification program is composed of a total of 8 personalized, one-hour face-to-face sessions. Participants will be encouraged to take on a moderate hypocaloric plan that cuts daily energy expenditure to encourage steady weight loss while preserving muscle mass. A protein intake of 1.5 g/kg of body weight per day is recommended. To optimize protein uptake, it's suggested that protein be distributed evenly across meals, aiming for 25-30 g per meal, inclusive of 2.5-2.8 g of leucine. Participants will also receive a guidebook, crafted through the Delphi method, to facilitate the adoption of these dietary modifications in their daily routines.
Behavioral: Exercise training — Participants will receive an 8-week program consisting of exercise training. It entails weekly group sessions, with each lasting an hour for 8 weeks. These sessions, designed for groups of approximately 10, will blend resistance and aerobic workouts to enhance muscle mass and strength while reducing fat in individuals with SO. Each session includes a 10-minute warm-up and cool-down, 20 minutes of resistance training using elastic bands, followed by a 20-minute brisk walking segment. Participants will also receive a YouTube link and a pamphlet describing the exercises, encouraging them to maintain at least 30 minutes of exercise five times a week during and beyond the supervised programme.
Behavioral: The EatWellLog App — Only participants in the M-health group will be instructed to use the EatWellLog app for daily diet self-management. This App supports participants with SO by providing a structured approach to managing a diet that encourages steady weight loss while maintaining muscle mass, in line with current nutritional recommendations for this demographic. The EatWellLog App has the following features: i) tracking participants' dietary habits by logging meals and snacks from a food list, ii) personalized online coaching and reminders by a multidisciplinary healthcare team, iii) participation of family caregivers through an interactive messaging function, iv) accessing health information via multiple channels, including animations, an at-a-glance display, and a reminder, and v) utilization of game elements, such as educational animations and video games to disseminate health and nutritional information related to SO.
  Arms: M-health group

SUMMARY:
Sarcopenic obesity, characterised by concurrent reduced muscle mass and excess body fat, affects 11% of older adults worldwide, rising to 23% in those over 75. Considering the negative synergistic impact on health, promoting muscle mass gains while reducing fat mass remains a significant challenge, necessitating urgent and effective intervention strategies for managing SO. Exercise and nutrition are the primary interventions recommended for SO.

This project aims to evaluate the effects of the EatWellLog App developed by the investigators' team for local older adults, in improving:

* their sarcopenic obesity status, measured by all four diagnostic criteria, including grip strength, muscle mass, physical performance and body fat mass (primary outcome), and,
* nutritional self-efficacy, nutritional status, dietary quality, health-related quality of life, and adherence to diet and exercise regimens (secondary outcomes), by enhancing the self-management abilities and longer-term adherence to daily diet management among participants in the M-health group using the App, compared to the control group.

The EatWellLog App, designed for older adults with SO, incorporating Klasnja and Pratt's five-strategy framework for mobile health (mHealth) applications development to facilitate health behavioural change. This App supports users with SO in managing daily diets that promote gradual weight loss and muscle mass preservation, adhering to the dietary regimen for this population.

Forty older adults with SO will be recruited from local community health centres and then randomized to either m-health or control groups. Both groups will receive an 8-week supervised programme separately. The programme consists of personalised dietary modification programme and group-based exercise training which have been tested and used in the investigators' pilot and General Research Fund (GRF) project. Additionally, only the m-health group will be instructed to use the App for daily diet self-management.

Participants will be assessed on a variety of outcomes immediately after the 8-week supervised programme (T1), which will be compared to the baseline (T0). To explore the possible long-term effects of the intervention, other measurements will be conducted at 3-(T2) and 6-(T3) months after the supervised programme, which will be compared with those conducted at T0.

DETAILED DESCRIPTION:
Sarcopenic obesity (SO), characterized by concurrent reduced muscle mass and excess body fat, affects 11% older adults worldwide, rising to 23% among those over 751. Older adults with reduced muscle mass are 1.95-2.62 times prone to obesity than those with normal muscle mass. This is due to shared etiological factors between sarcopenia and obesity such as sedentary habits and aging-related biological shifts, including decreased anabolic hormones, increased insulin resistance, and escalated oxidative stress. The combination of sarcopenia and obesity has a compounding negative impact on health, raising the likelihood of knee and hip osteoarthritis, which leads to reduced physical capabilities, as well as increasing the risk of cardio-metabolic diseases, institutionalized, and death, exceeding the risks of sarcopenia or obesity alone.

Addressing SO effectively to promote muscle mass gains while reducing fat mass remains a significant challenge, necessitating urgent and effective intervention strategies. Currently, exercise and nutrition interventions, are the most commonly recommended interventions.

Exercise and Nutrition Interventions for SO A recent systematic review of 11 trials with 440 SO participants showed that resistance training twice weekly for 20 minutes over a minimum of 8 weeks effectively enhances body composition, muscle strength, and gait speed. Furthermore, evidence suggested that combining aerobic and resistance training with increased protein intake is more effective in reducing body fat than resistance training alone but had no effects on muscle mass and strength. Another systematic review of eight trials with 605 SO participants found that resistance training alone could increase muscle strength. To also improve physical functions (i.e., gait speed and grip strength), exercise combining aerobic and resistance training with dietary supplements seems to have more promising results. The findings in a recent umbrella review of meta-analyses concluded that exercise interventions (either resistance training or combined resistance and aerobic exercise) are beneficial for body composition and physical performance in older adults with SO. However, the added value of exercise with nutrition interventions (either protein supplement and dietary modifications) produces inconsistent results.

Adequate protein intake is vital for muscle building, and calorie restriction is effective at reducing fat mass. Thus, nutrition is a critical factor in the onset and progression of SO, although the evidence for nutrition interventions in reserving SO demonstrated inconsistent effects, especially regarding muscle mass and strength. When implementing a weight loss diet for individuals with SO, it is important to balance fat reduction with muscle mass preservation by ensure adequate protein intake to prevent exacerbating muscle loss. Evidence suggests that the source of protein is crucial for muscle retention, specifically for animal-based proteins, which are high in leucine, may be more effective in preserving muscle mass during weight loss and in maintaining physical function. While nutritional supplements are commonly used to increase protein intake, their effects on SO remain inconsistent and may cause side effects such as digestive issues, interact with certain medications, dehydration, liver and renal damage, bloating, and calcium loss. The investigators advocates for an unhealthy diet incorporating a full spectrum of nutrients from whole foods, in line with the Dietary Guidelines for Americans, 2020-2025, as the preferred approach over supplements for those with sarcopenic obesity. Modifying daily dietary habits of individuals with SO may provide more sustainable benefits than merely adding supplements to their diet.

A recent systematic review examining nutrition interventions in managing sarcopenic obesity analysed nine studies but only two assessed the impact of dietary modifications on protein intake among older adults with SO. The first randomized controlled trial (RCT) assessed the impact of a low-calorie diet with normal (0.8 g/kg body weight/day) versus high protein intake (1.2 g/kg body weight/day) over three months in 104 older women with SO. The study found muscle mass decreased in the normal protein group concurrent with fat loss, while the high protein group saw muscle mass preservation. The second pilot RCT involving 18 women compared a low-calorie diet with placebo to one with high protein (1.2-1.4 g/kg body weight/day) over four months. Significant muscle strength gains were noted in the high protein group, though changes in muscle mass were not significantly different between the two groups. While the findings in these two trials provided preliminary evidence that hypocaloric diet and high protein intake may be necessary for managing SO, particularly for preserving mass muscle and strength. These studies, however, had limitations such as broad inclusion criteria for sarcopenic obesity, lacking a standardized diagnostic protocol, insufficient data on dietary adherence, and opaque details regarding randomization and intervention specifics. More rigorous research is needed to investigate the impact of diet modification on sarcopenic obesity.

Conventional dietary modification intervention that relies on face-to-face consultation and monitoring, faced lots of challenges which included participants' poor compliance to the recommended dietary regimen, high attrition, time constraints and manpower. Those were major threats to the viability of the study leading to inconsistent treatment effects. In addition, the therapeutic effect may gradually reduces after the completion of the dietary training program. Additionally, the therapeutic effect may gradually reduce after the completion of the dietary program.

Rationale for developing a m-health based intervention for SO Systematic reviews found that m-health dietary intervention, with appropriate behaviour change techniques, can achieve dietary behaviour change across a range of chronic illnesses, such as obesity, metabolic syndrome, cardiovascular disease with relatively low attrition rates. To the best of the knowledge, there are no studies evaluating the effects of m-health dietary interventions on SO. The success of m-health interventions in other chronic conditions could potentially be adapted to improve health behaviors in patients with SO.

Aims and Hypotheses to be Tested.

The study aims to evaluate the effects of the EatWellLog App (hereafter referred to as "the App"), designed by the investigators' team to address the needs of local older adults, in improving:

* their sarcopenic obesity status, measured by all four diagnostic criteria, including grip strength, muscle mass, physical performance and body fat mass (primary outcome), and,
* nutritional self-efficacy, nutritional status, dietary quality, health-related quality of life, and adherence to diet and exercise regimens (secondary outcomes), by enhancing the self-management abilities and longer-term adherence to daily diet management among participants in the M-health group using the App, compared to the control group.

It is hypothesised that the App users will demonstrate significant and sustained improvements in SO status and secondary outcomes immediately after the supervised nutrition and exercise programme and at 3-and 6-month follow ups, compared to the control group who receive the same supervised programme without the App.

The investigators will also explore users' experience with the App by focus groups with all participants in the M-health group, 6-8 per group, to understand their experience of using the App. Additionally, the investigators will analyse the App usage data including session duration, frequency, feature utilisation, and retention rates, at the 3-month and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or above, and living in the community;
* Having SO according to the Asian Working Group for Sarcopenia (AWGS) and the World Health Organization (WHO)'s obesity criteria for Asians:

  1. Early-stage sarcopenia indicated by fulfilment of one of the following criteria; handgrip strength <28 kg (men) and <18 kg (women); appendicular skeletal muscle mass (ASM)/ height2 <7 kg/m2 (men) and <5.7 kg/m2 (women), or SPPB score of <9; Short Physical Performance Battery (SPPB) score of <9,
  2. Obesity indicated by BMI ≥25 kg/m2, waist circumference ≥90 cm (men) and ≥80 cm (women), or body fat >30%;
* Own a smartphone with internet access; and
* Proficiency in communicating, reading, and writing in Chinese, and without major hearing and vision impairments to ensure that comprehension of our instructions.

Exclusion Criteria:

* Individuals with diseases impacting digestion or food consumption, including severe cardiac/ pulmonary/ renal diseases, diabetes, cancer, or autoimmune disorders;
* Those on medications affecting eating habits, digestion, or metabolism, such as weight loss drugs;
* Persons with alcohol use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), potentially hindering dietary behaviour changes;
* Those with medical implants like pacemakers that could be disrupted by the bioelectric impedance analysis (BIA's) low-level electrical currents.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes of muscle strength | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Handgrip strength (kg) will be measured by using the hand dynamometer.
Changes of muscle mass | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Muscle mass (kg) will be measured by using bioelectrical impedance analysis.
Changes of body mass index | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The weight and height will be combined to report BMI in kg/m^2.
Changes of waist circumference | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Waist circumference was taken as the minimum circumference between the umbilicus and xiphoid process and measured to the nearest 0.5 cm.
Changes of fat mass | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Fat mass (kg) will be measured by using bioelectrical impedance analysis.
The Short Physical Performance Battery (SPPB) scale | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The Short Physical Performance Battery (SPPB) scale will be used to measure physical function, which is a well-established tool for monitoring function in older people, which contains three kinds of assessments: stand for 10 seconds with feet in 3 different positions, 3-meter or 4-meter walking speed test, and time to rise from a chair for five times. The scores of SPPB range from 0 (worst performance) to 12 (best performance). The minimum and maximum values are 0 and 10 respectively. Higher scores mean a better performance.

SECONDARY OUTCOMES:
Mini Nutritional Assessment (MNA) Short-form | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Participants' nutritional status will be assessed through the Mini Nutritional Assessment (MNA). It is a simple and quick tool for assessing older people who are malnourished or at risk of malnutrition. The MNA Short-form contains 6 items. Questions are weighted, 2-3 points per item. Scores are categorised as 0-7 (malnourished), 8-11 (at risk of malnutrition), 12-14 (normal nutritional status). The minimum and maximum values are 0 and 14 respectively. Higher scores mean a better nutritional status.
Health Action Process Approach (HAPA) Nutrition Self-efficacy Scale | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The nutrition self-efficacy scale is one part of the Health-Specific Self-efficacy Scale. The nutritional self-efficacy scale is a 5-item scale, and each item is rated on 4-point likert scale from 1= very uncertain, 2=rather uncertain, 3=rather certain, 4=very certain. Higher score means higher self-efficacy. The minimum and maximum values are 0 and 20 respectively. Higher scores mean a higher self-efficacy.
Dietary Quality Index-International (DQI-I) | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The DQI-I will be used to estimate the dietary quality of participants. It is a well-used questionnaire without being affected by culture. The total scores range from 0 to 100, with a higher score representing better diet quality. The minimum and maximum values are 0 and 100 respectively. Higher scores mean a better diet quality.
EuroQoL 5D (EQ-5D) | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The EQ-5D comprises five dimensions of health: mobility, self-care, usual activities, pain / discomfort, and anxiety/depression. Each of them has three response categories: no, some, or extreme problems, and a 0-100 points visual analogue scale (EQ VAS). The ratings from the five categories can be transformed into a utility index score by utilizing the scores derived from the preference weights of the general population in Hong Kong. The utility score generally ranges from less than 0 to 1. A higher score indicates higher health utility. The EQ VAS ranges from 0 to 100, with higher scores indicate better imaginable health.
Diet Adherence | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  The adherence to protein intake will be analyzed by a software program "Food Processor®". If any participant forgets to keep the dietary record, the 7-day food recall method will be used by the experimental group facilitator to check the participant's food intake, an approach commonly used in nutritional studies.
Exercise Adherence | Change from baseline to 8 weeks, 3 months, and 6 months after completing the program
  Assessed based on the participants' self-reports on their overall adherence to the exercise regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Justina Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the information of all participants will be replaced by reference codes. The data collected will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 7 years after the completion of this research.

REFERENCES:
- [Background] Gao Q, Mei F, Shang Y, Hu K, Chen F, Zhao L, Ma B. Global prevalence of sarcopenic obesity in older adults: A systematic review and meta-analysis. Clin Nutr. 2021 Jul;40(7):4633-4641. doi: 10.1016/j.clnu.2021.06.009. Epub 2021 Jun 21. PMID 34229269
- [Background] Stenholm S, Harris TB, Rantanen T, Visser M, Kritchevsky SB, Ferrucci L. Sarcopenic obesity: definition, cause and consequences. Curr Opin Clin Nutr Metab Care. 2008 Nov;11(6):693-700. doi: 10.1097/MCO.0b013e328312c37d. PMID 18827572
- [Background] Polyzos SA, Margioris AN. Sarcopenic obesity. Hormones (Athens). 2018 Sep;17(3):321-331. doi: 10.1007/s42000-018-0049-x. Epub 2018 Jul 16. PMID 30014320
- [Background] Kob R, Bollheimer LC, Bertsch T, Fellner C, Djukic M, Sieber CC, Fischer BE. Sarcopenic obesity: molecular clues to a better understanding of its pathogenesis? Biogerontology. 2015 Feb;16(1):15-29. doi: 10.1007/s10522-014-9539-7. Epub 2014 Nov 7. PMID 25376109
- [Background] Nakano R, Takebe N, Ono M, Hangai M, Nakagawa R, Yashiro S, Murai T, Nagasawa K, Takahashi Y, Satoh J, Ishigaki Y. Involvement of oxidative stress in atherosclerosis development in subjects with sarcopenic obesity. Obes Sci Pract. 2017 Jan 27;3(2):212-218. doi: 10.1002/osp4.97. eCollection 2017 Jun. PMID 28702214
- [Background] Godziuk K, Prado CM, Woodhouse LJ, Forhan M. The impact of sarcopenic obesity on knee and hip osteoarthritis: a scoping review. BMC Musculoskelet Disord. 2018 Jul 28;19(1):271. doi: 10.1186/s12891-018-2175-7. PMID 30055599
- [Background] Nezameddin R, Itani L, Kreidieh D, El Masri D, Tannir H, El Ghoch M. Understanding Sarcopenic Obesity in Terms of Definition and Health Consequences: A Clinical Review. Curr Diabetes Rev. 2020;16(9):957-961. doi: 10.2174/1573399816666200109091449. PMID 31916519
- [Background] Alexandre TDS, Scholes S, Ferreira Santos JL, Duarte YAO, de Oliveira C. The combination of dynapenia and abdominal obesity as a risk factor for worse trajectories of IADL disability among older adults. Clin Nutr. 2018 Dec;37(6 Pt A):2045-2053. doi: 10.1016/j.clnu.2017.09.018. Epub 2017 Oct 2. PMID 29033231
- [Background] Reiter L, Bauer S, Traxler M, Schoufour JD, Weijs PJM, Cruz-Jentoft A, Topinkova E, Eglseer D. Effects of Nutrition and Exercise Interventions on Persons with Sarcopenic Obesity: An Umbrella Review of Meta-Analyses of Randomised Controlled Trials. Curr Obes Rep. 2023 Sep;12(3):250-263. doi: 10.1007/s13679-023-00509-0. Epub 2023 May 30. PMID 37249818
- [Background] Eglseer D, Traxler M, Schoufour JD, Weijs PJM, Voortman T, Boirie Y, Cruz-Jentoft AJ, Reiter L, Bauer S; SO-NUTS Consortium. Nutritional and exercise interventions in individuals with sarcopenic obesity around retirement age: a systematic review and meta-analysis. Nutr Rev. 2023 Aug 10;81(9):1077-1090. doi: 10.1093/nutrit/nuad007. PMID 36882046
- [Background] Hita-Contreras F, Bueno-Notivol J, Martinez-Amat A, Cruz-Diaz D, Hernandez AV, Perez-Lopez FR. Effect of exercise alone or combined with dietary supplements on anthropometric and physical performance measures in community-dwelling elderly people with sarcopenic obesity: A meta-analysis of randomized controlled trials. Maturitas. 2018 Oct;116:24-35. doi: 10.1016/j.maturitas.2018.07.007. Epub 2018 Jul 19. PMID 30244776
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. Aging is associated with diminished accretion of muscle proteins after the ingestion of a small bolus of essential amino acids. Am J Clin Nutr. 2005 Nov;82(5):1065-73. doi: 10.1093/ajcn/82.5.1065. PMID 16280440
- [Background] Mathus-Vliegen EM; Obesity Management Task Force of the European Association for the Study of Obesity. Prevalence, pathophysiology, health consequences and treatment options of obesity in the elderly: a guideline. Obes Facts. 2012;5(3):460-83. doi: 10.1159/000341193. Epub 2012 Jun 30. PMID 22797374
- [Background] Abiri B, Hosseinpanah F, Seifi Z, Amini S, Valizadeh M. The Implication of Nutrition on the Prevention and Improvement of Age-Related Sarcopenic Obesity: A Systematic Review. J Nutr Health Aging. 2023;27(10):842-852. doi: 10.1007/s12603-023-1986-x. PMID 37960907
- [Background] Trouwborst I, Verreijen A, Memelink R, Massanet P, Boirie Y, Weijs P, Tieland M. Exercise and Nutrition Strategies to Counteract Sarcopenic Obesity. Nutrients. 2018 May 12;10(5):605. doi: 10.3390/nu10050605. PMID 29757230
- [Background] Sammarco R, Marra M, Di Guglielmo ML, Naccarato M, Contaldo F, Poggiogalle E, Donini LM, Pasanisi F. Evaluation of Hypocaloric Diet With Protein Supplementation in Middle-Aged Sarcopenic Obese Women: A Pilot Study. Obes Facts. 2017;10(3):160-167. doi: 10.1159/000468153. Epub 2017 May 20. PMID 28528340
- [Background] Rehman SU, Ali R, Zhang H, Zafar MH, Wang M. Research progress in the role and mechanism of Leucine in regulating animal growth and development. Front Physiol. 2023 Nov 17;14:1252089. doi: 10.3389/fphys.2023.1252089. eCollection 2023. PMID 38046946
- [Background] Hsu KJ, Liao CD, Tsai MW, Chen CN. Effects of Exercise and Nutritional Intervention on Body Composition, Metabolic Health, and Physical Performance in Adults with Sarcopenic Obesity: A Meta-Analysis. Nutrients. 2019 Sep 9;11(9):2163. doi: 10.3390/nu11092163. PMID 31505890
- [Background] Schaafsma G. Safety of protein hydrolysates, fractions thereof and bioactive peptides in human nutrition. Eur J Clin Nutr. 2009 Oct;63(10):1161-8. doi: 10.1038/ejcn.2009.56. Epub 2009 Jul 22. PMID 19623200
- [Background] U.S. Department of Agriculture & U.S. Department of Health and Human Services. Dietary Guidelines for Americans, 2020-2025. December 2020. Accessed 1 Feb 2024. https://www.dietaryguidelines.gov/sites/default/files/2020-12/Dietary_Guidelines_for_Americans_2020-2025.pdf
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Background] Muscariello E, Nasti G, Siervo M, Di Maro M, Lapi D, D'Addio G, Colantuoni A. Dietary protein intake in sarcopenic obese older women. Clin Interv Aging. 2016 Feb 5;11:133-40. doi: 10.2147/CIA.S96017. eCollection 2016. PMID 26917955
- [Background] Yin YH, Liu JYW, Valimaki M. Effectiveness of non-pharmacological interventions on the management of sarcopenic obesity: A systematic review and meta-analysis. Exp Gerontol. 2020 Jul 1;135:110937. doi: 10.1016/j.exger.2020.110937. Epub 2020 Mar 30. PMID 32240820
- [Background] Crichton GE, Howe PR, Buckley JD, Coates AM, Murphy KJ, Bryan J. Long-term dietary intervention trials: critical issues and challenges. Trials. 2012 Jul 20;13:111. doi: 10.1186/1745-6215-13-111. PMID 22812577
- [Background] Burgess E, Hassmen P, Pumpa KL. Determinants of adherence to lifestyle intervention in adults with obesity: a systematic review. Clin Obes. 2017 Jun;7(3):123-135. doi: 10.1111/cob.12183. Epub 2017 Mar 15. PMID 28296261
- [Background] Young C, Campolonghi S, Ponsonby S, Dawson SL, O'Neil A, Kay-Lambkin F, McNaughton SA, Berk M, Jacka FN. Supporting Engagement, Adherence, and Behavior Change in Online Dietary Interventions. J Nutr Educ Behav. 2019 Jun;51(6):719-739. doi: 10.1016/j.jneb.2019.03.006. Epub 2019 Apr 27. PMID 31036500
- [Background] Paddon-Jones D, Leidy H. Dietary protein and muscle in older persons. Curr Opin Clin Nutr Metab Care. 2014 Jan;17(1):5-11. doi: 10.1097/MCO.0000000000000011. PMID 24310053
- [Background] Eyles HC, Mhurchu CN. Does tailoring make a difference? A systematic review of the long-term effectiveness of tailored nutrition education for adults. Nutr Rev. 2009 Aug;67(8):464-80. doi: 10.1111/j.1753-4887.2009.00219.x. PMID 19674343
- [Background] Klasnja P, Pratt W. Healthcare in the pocket: mapping the space of mobile-phone health interventions. J Biomed Inform. 2012 Feb;45(1):184-98. doi: 10.1016/j.jbi.2011.08.017. Epub 2011 Sep 9. PMID 21925288
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] World Health Organization. The Asia-Pacific perspective: redefining obesity and its treatment. February 2000. Accessed 10 Jan 2024. https://iris.who.int/bitstream/handle/10665/206936/0957708211_eng.pdf
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Liu P, Ma F, Lou H, Zhu Y. Utility of obesity indices in screening Chinese postmenopausal women for metabolic syndrome. Menopause. 2014 May;21(5):509-14. doi: 10.1097/GME.0b013e3182a170be. PMID 23963310
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). American Psychiatric Association.
- [Background] InBody. (2024). InBody S10. https://inbodyusa.com/products/inbodyS10/
- [Background] Yin YH, Liu JYW, Valimaki M. Dietary behaviour change intervention for managing sarcopenic obesity among community-dwelling older people: a pilot randomised controlled trial. BMC Geriatr. 2023 Sep 26;23(1):597. doi: 10.1186/s12877-023-04327-w. PMID 37752447
- [Background] Liu J ZY, Lo K, et al,. Effects of an Individualized Dietary Behavioural Change (IDBC) Programme and Exercise Training in combination or separately on managing sarcopenic obesity in community-dwelling older adults: A Randomized Controlled Trial (ongoing GRF project).
- [Background] Liu, JYW. (2023). Things to know about Sarcopenic Obesity: A dietary guide for older adults with muscle loss and excessive body fat. School of Nursing, The Hong Kong Polytechnic University.
- [Background] Kraus WE, Bhapkar M, Huffman KM, Pieper CF, Krupa Das S, Redman LM, Villareal DT, Rochon J, Roberts SB, Ravussin E, Holloszy JO, Fontana L; CALERIE Investigators. 2 years of calorie restriction and cardiometabolic risk (CALERIE): exploratory outcomes of a multicentre, phase 2, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):673-683. doi: 10.1016/S2213-8587(19)30151-2. Epub 2019 Jul 11. PMID 31303390
- [Background] Bauer J, Biolo G, Cederholm T, Cesari M, Cruz-Jentoft AJ, Morley JE, Phillips S, Sieber C, Stehle P, Teta D, Visvanathan R, Volpi E, Boirie Y. Evidence-based recommendations for optimal dietary protein intake in older people: a position paper from the PROT-AGE Study Group. J Am Med Dir Assoc. 2013 Aug;14(8):542-59. doi: 10.1016/j.jamda.2013.05.021. Epub 2013 Jul 16. PMID 23867520
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] U.S. Department of Agriculture, Agricultural Research Service. FoodData Central, 2019. fdc.nal.usda.gov.
- [Background] Guerra RS, Amaral TF. Comparison of hand dynamometers in elderly people. J Nutr Health Aging. 2009 Dec;13(10):907-12. doi: 10.1007/s12603-009-0250-3. PMID 19924352
- [Background] Schwarzer, R., & Renner, B. (2009). Health-specific self-efficacy scales. Freie Universität Berlin, 14, 2009.
- [Background] He, X. Y., & Liu, X. Q. (2010). Evaluation of reliability and validity of Mini-nutritional assessment and Chinese nutrition screen. Nurs J Chin People's Liberation Army, 27, 894-6.
- [Background] Kim S, Haines PS, Siega-Riz AM, Popkin BM. The Diet Quality Index-International (DQI-I) provides an effective tool for cross-national comparison of diet quality as illustrated by China and the United States. J Nutr. 2003 Nov;133(11):3476-84. doi: 10.1093/jn/133.11.3476. PMID 14608061
- [Background] Yang YJ, Kim MK, Hwang SH, Ahn Y, Shim JE, Kim DH. Relative validities of 3-day food records and the food frequency questionnaire. Nutr Res Pract. 2010 Apr;4(2):142-8. doi: 10.4162/nrp.2010.4.2.142. Epub 2010 Apr 28. PMID 20461203
- [Background] Wang HM, Patrick DL, Edwards TC, Skalicky AM, Zeng HY, Gu WW. Validation of the EQ-5D in a general population sample in urban China. Qual Life Res. 2012 Feb;21(1):155-60. doi: 10.1007/s11136-011-9915-6. Epub 2011 Apr 20. PMID 21505881
- [Background] Food Processor® software [Computer software]. (2023). Retrieved from https://esha.com/products/food-processor/
- [Background] Rafique, H., Almagrabi, A. O., Shamim, A., Anwar, F., & Bashir, A. K. (2020). Investigating the acceptance of mobile library applications with an extended technology acceptance model (TAM). Computers & Education, 145, 103732.
- [Background] Krippendorff K. (2018). Content analysis: An introduction to its methodology. SAGE Publications, Inc.
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063

DOCUMENTS (1):
  • Informed Consent Form (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT06360432/ICF_000.pdf